CLINICAL TRIAL: NCT03718104
Title: Safety, Efficacy, Pharmacokinetics, and Pharmacogenomics of Extended-Release Naltrexone in Pregnant Women
Brief Title: MOM NEST Study: Maternal Opioid Medication: Naltrexone Efficacy Study
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: University of North Carolina (Other); University of California, San Diego (Other); Boston University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-37773; R01HD096798-01 (NIH)
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Opioid-use Disorder; Neonatal Abstinence Syndrome; Pregnancy, High Risk; Alcohol Use Disorder
Keywords: naltrexone; buprenorphine/naloxone; maternal relapse; retention in care; pharmacokinetics; pharmacogenetics
MeSH Terms: conditions — Opioid-Related Disorders; Neonatal Abstinence Syndrome; Alcoholism | interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal and infant blood and urine samples for naltrexone pharmacokinetics
  * Cord blood for naltrexone pharmacokinetics
  * Breast milk for naltrexone levels
  * Maternal blood, saliva, and placental tissue for genotyping and DNA methylation
  * Maternal and infant samples for cortisol levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Naltrexone: Pregnant women with opioid use disorder on prescribed oral or extended-release naltrexone and their infants. Biospecimens collected from this group will undergo pharmacokinetic analysis, genetic and epigenetic analysis, and breast milk analysis. This group will also receive safety and efficacy interventions.
  Interventions: Other: Pharmacokinetic analysis; Other: Safety and Efficacy; Genetic: Genetic and epigenetic analysis; Other: Breast milk analysis
- Buprenorphine/Naloxone: Pregnant women with opioid use disorder on prescribed buprenorphine/naloxone and their infants. Biospecimens collected from this group will undergo genetic and epigenetic analysis and the group will also receive safety and efficacy interventions.
  Interventions: Other: Safety and Efficacy; Genetic: Genetic and epigenetic analysis
- Naltrexone - alcohol use disorder: Pregnant women with alcohol use disorder on prescribed naltrexone (oral or extended-release) and their infants. Biospecimens collected from this group will undergo pharmacokinetic analysis, genetic and epigenetic analysis, and breast milk analysis. This exploratory group will also receive safety and efficacy interventions.
  Interventions: Other: Pharmacokinetic analysis; Genetic: Genetic and epigenetic analysis; Other: Breast milk analysis

INTERVENTIONS:
Other: Pharmacokinetic analysis — Pharmacokinetic analysis of maternal blood, maternal urine, cord blood, infant blood and urine for dyads in the naltrexone group at various time points in the pregnancy, at delivery, and 4 weeks postpartum.
  Groups: Naltrexone; Naltrexone - alcohol use disorder
Other: Safety and Efficacy — Examination of the safety and efficacy of naltrexone and comparison of outcomes with the buprenorphine/naloxone cohort. Outcomes examined will include: 1) maternal outcomes (relapse, retention in care, preterm labor); 2) fetal outcomes (growth, fetal anomalies, fetal distress, cortisol levels); and 3) infant outcomes (NAS, growth, neurodevelopment via NNNS exam at 4 weeks and Bayley exam at 12 months of age).
  Groups: Buprenorphine/Naloxone; Naltrexone
Genetic: Genetic and epigenetic analysis — Maternal blood and saliva DNA samples will be genotyped for single nucleotide polymorphisms in the mu opioid receptor gene (OPRM1) to look for associations with effectiveness of NTX and BPH. In addition, DNA methylation levels in the OPRM1 promoter within maternal and infant saliva and placenta at delivery and 4 weeks postpartum will be examined. Lastly, we will compare genome-wide DNA methylation levels at delivery and 4 weeks postpartum in mother-infant dyads.
Other: Breast milk analysis — Mothers in the naltrexone group will have their breast milk analyzed at 4 weeks post-delivery for naltrexone levels, with corresponding maternal and infant plasma levels.
  Groups: Naltrexone; Naltrexone - alcohol use disorder

SUMMARY:
This is a multi-center prospective comparative cohort study examining the safety, efficacy, pharmacokinetics, and pharmacogenomics of naltrexone for pregnant women with opioid use disorder. Pregnancy, delivery, and maternal and infant outcomes to 12 months post-delivery will be examined and compared with a cohort treated with buprenorphine/naloxone.

DETAILED DESCRIPTION:
Fifty pregnant women stabilized pre-pregnancy on oral or extended-release naltrexone (XR-NTX) and 50 comparison women on buprenorphine/naloxone (BPH) from Boston Medical Center and the University of North Carolina will be enrolled in this multi-center prospective comparative cohort study. The specific aims of this project are: 1) Safety and Efficacy: To compare maternal outcomes (safety, relapse, retention in care), fetal outcomes (growth, fetal distress), and infant outcomes (neonatal abstinence syndrome, growth, neurodevelopment) during pregnancy until 12 months post- delivery; An exploratory part of this aim is to collect safety and efficacy data on women receiving NTX for alcohol use disorder (AUD). We will collect maternal, fetal and infant outcomes related to prenatal alcohol exposure. 2) Pharmacokinetics: To determine the pharmacokinetics of NTX in pregnant and postpartum women; 3) Genetics and Epigenetics: To examine the association between genetic variants and epigenetic modification in the mu-opioid receptor (OPRM1) gene, as well as global DNA methylation changes after treatment with NTX and BPH within the mother, placenta, and infant; and 4) Breast milk: To measure breast milk concentrations of NTX and corresponding infant relative dose to determine safety for lactating women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 6 - 30 6/7 weeks gestation, receiving prenatal care at Boston Medical Center (BMC) or the University of North Carolina (UNC)
* Plan to deliver infant at BMC or UNC
* Diagnosis of opioid use disorder (OUD) or alcohol use disorder (AUD) in the current pregnancy on prescribed oral or extended-release naltrexone; or buprenorphine/naloxone for the treatment of OUD
* English speaking
* Singleton pregnancy

Exclusion Criteria:

* OUD on prescribed methadone, or no maintenance medication
* OUD on Subutex formulation of buprenorphine
* Severe psychiatric illness or cognitively impairing ability to provide informed consent
* Current maternal incarceration
* Women who present for care >31 0/7 weeks
* Multiple gestation pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women with opioid use disorder or alcohol use disorder on prescribed naltrexone, or those with opioid use disorder on buprenorphine/naloxone and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Maternal drug use relapse | up to 12 months post-delivery
  Maternal relapse of illicit and/or unprescribed drug use from maternal/provider report and or from urine toxicology testing at any point during the pregnancy and up to 12 months after delivery

SECONDARY OUTCOMES:
Naltrexone side effects or adverse events | up to 12 months post-delivery
  Number and type of side effects or adverse events such as injection site reactions, gastrointestinal upset, syncope, headaches, or dizziness reported by participant or provider
Fetal heart rate monitoring from NST | 27- 41 weeks gestation
  Mean fetal heart rate (FHR), FHR variability, and episodic accelerations of FHR (count) from each routine care non-stress test (NST) in the third trimesters.
Biophysical profile score calculated from NST | 27 - 41 weeks gestation
  The biophysical profile uses electronic fetal heart rate monitoring to examine the fetus. There are five components measured during the biophysical examination (fetal breathing movements, gross body movement, fetal tone, amninotic fluid volume and whether the NST is reactive or nonreactive. A score of 2 points is given for each component The points are then added for a possible maximum score of 10. The test is continued until all criteria are met or 30 minutes have elapsed. HIgher scores are more favorable.
Maternal hair cortisol levels | Birth and 4 weeks post-delivery
  Hair cortisol levels will be obtained from maternal hair samples obtained at birth and 4 weeks after delivery, and compared between the naltrexone and buprenorphine groups. Higher hair cortisol levels in the mother may indicate exposure to higher levels of stress over the preceding 3 months period.
Infant hair cortisol levels | Birth and 4 weeks post-delivery
  Hair cortisol levels will be obtained from infant hair samples obtained at birth and 4 weeks after delivery, and compared between the naltrexone and buprenorphine groups. Higher hair cortisol levels in the infant may indicate exposure to higher levels of stress over the preceding 3 months period.
Fetal growth based on ultrasound measurements | 18 - 41 weeks gestation
  Fetal growth will be assessed at the time of routine growth scans at 18-20, and then q4 weeks until delivery. Fetal size will be compared to Intergrowth standards to produce z-scores and SGA (<10%ile) for averaged 2nd and 3rd trimester measurements.
Congenital fetal anomalies by ultrasound | 18 - 41 weeks gestation
  Fetal, placental, or amniotic fluid anomalies identified during routine ultrasounds in the second and third trimesters will be documented.
Congenital anomalies by physical examination | Birth
  Infants will be routinely assessed at birth during the physical examination for any external anomalies.
Diagnosis of Neonatal Abstinence Syndrome (NAS) | From birth to 30 days
  NAS diagnosis will be based on opioid withdrawal signs and symptoms in the infant after delivery as assessed by NAS withdrawal scores (either the Finnegan score or the via the ESC (Eat, Sleep, Console) assessment tool. The Finnegan scale assesses 21 of the most common signs of neonatal drug withdrawal syndrome and is scored on the basis of pathological significance and severity of the adverse symptoms, which sometimes requires pharmacological treatment. Measurements are performed every 4 hours, typically with 2-3 consecutive scores that are equal to or greater than 8, or 1-2 scores of 12 or greater, pharmacologic treatment for withdrawal is started. For the ESC assessment, clinicians assess whether or not the infant has poor feeding, is unable to sleep for at least 1 hour after feeding, and is consolable (rating of 1-3) due to symptoms of opioid withdrawal. Poor feeding, sleeping, or consolability triggers a huddle and possible start of pharmacologic treatment.
Infant need for pharmacologic treatment | From birth to 30 days
  The need for pharmacologic treatment will be recorded as Y/N as will the need for adjunctive agents.
Infant need for adjunctive agent | From birth to 30 days
  The need for adjunctive agents will be recorded as Y/N
Infant opioid replacement pharmacologic treatment | From birth to 30 days
  The total mgs of morphine/methadone needed for pharmacologic treatment and the total number of total opioid treatment days will be obtained from the birth hospitalization medical records.
Infant birth hospitalization length of stay | From birth to 30 days
  Number of continuous days infant hospitalized after birth.
Infant weight | Birth, 4 weeks, and 12 months
  Growth parameters of infant weight in grams will be obtained by the clinician at birth, 4 weeks, and 12 months at each study visit. Percentiles will be calculated.
Infant length | Birth, 4 weeks, and 12 months
  Growth parameters of infant length measured by the clinician in cm will be obtained at birth, 4 weeks, and 12 months at each study visit. Percentiles will be calculated.
Infant head circumference | Birth, 4 weeks, and 12 months
  Growth parameters of infant head circumference in cm will be obtained by the clinician at birth, 4 weeks, and 12 months at each study visit. Percentiles will be calculated.
Infant neurobehavior-function assessed by the NNNS | 4 weeks of age
  The NICU Network Neurobehavioral Scale (NNNS) is a comprehensive assessment of both neurologic integrity and behavioral functioning, including signs of stress. It assesses the full range of infant neurobehavioral performance (orientation to auditory and visual stimuli); infant stress (color changes, tremors, startles), neurologic functioning (reflexes, tone); some features of gestational age; self-soothing capacities; states and their organization. The 13 summary scores (i.e., orientation, habituation, hypertonicity, hypotonicity, excitability, arousal, lethargy, non-optimal reflexes, asymmetric reflexes, stress, self-regulation, quality of movement, handling) are typically used to summarize a clinical examination .
Infant neurodevelopment assessed by Bayley III | 12 months of age
  The Bayley III is a standard series of measurements used to assess the development of infants and toddlers, ages 1-42 months. It has 5 scales, 3 administered with child interaction - cognitive, motor, language, and 2 with parent questionnaires- social-emotional, adaptive behavior. A developmental quotient (DQ) is derived from the results.
Pharmacokinetic analysis of maternal naltrexone levels | 2nd trimester, 3rd trimester, delivery, 2-4 days after delivery, 4 weeks post-delivery
  Naltrexone levels from maternal blood and plasma will be obtained at regular intervals for pharmacokinetic analysis.
Pharmacokinetic analysis of infant naltrexone levels | Delivery, 2-4 days after delivery, 4 weeks post-delivery
  Naltrexone levels from infant blood and plasma will be obtained at regular intervals for pharmacokinetic analysis.

OTHER OUTCOMES:
Maternal DNA methylation profile | 36 weeks gestation
  Mothers will have a genome wide methylation profile at 36 weeks gestation from a blood sample.
Mu opioid receptor (OPRM1) gene single nucleotide (SNP) genotype | 36 weeks gestation
  Mothers will be genotyped for the ORPM1 A118G SNP at 36 weeks gestation from a blood sample to see if genotype is associated with treatment response and risk for relapse.
Maternal saliva OPRM1 methylation status | Birth, 4 weeks postpartum
  Mothers will have their OPRM1 methylation status examined via saliva samples to see if OPRM1 methylation is altered by maternal treatment.
Infant saliva OPRM1 methylation status | Birth, 4 weeks postpartum
  Infants will have their OPRM1 methylation status examined via saliva samples at to see if OPRM1 methylation is altered by maternal treatment.
Breast milk naltrexone level | 4 weeks postpartum
  Naltrexone levels will be measured from the breast milk of breastfeeding mothers who are on naltrexone.
Retention in addiction treatment | up to 12 months post-delivery
  Length of time mother continues medication assisted treatment (MAT) from provider or participant report
Maternal healthcare utilization | up to 12 months post-delivery
  Data on maternal healthcare utilization, including emergency room visits, primary care visits, and re-hospitalizations will be collected.
Infant healthcare utilization | up to 12 months post-delivery
  Data on infant healthcare utilization, including emergency room visits, primary care visits, and re-hospitalizations will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Elisha Wachman, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - University of North Carolina Chapel Hill, Carrboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones HE, Chisolm MS, Jansson LM, Terplan M. Naltrexone in the treatment of opioid-dependent pregnant women: the case for a considered and measured approach to research. Addiction. 2013 Feb;108(2):233-47. doi: 10.1111/j.1360-0443.2012.03811.x. Epub 2012 Apr 4. PMID 22471668
- [Background] Saia KA, Schiff D, Wachman EM, Mehta P, Vilkins A, Sia M, Price J, Samura T, DeAngelis J, Jackson CV, Emmer SF, Shaw D, Bagley S. Caring for Pregnant Women with Opioid Use Disorder in the USA: Expanding and Improving Treatment. Curr Obstet Gynecol Rep. 2016;5(3):257-263. doi: 10.1007/s13669-016-0168-9. Epub 2016 Jul 1. PMID 27563497
- [Background] Wachman EM, Saia K, Miller M, Valle E, Shrestha H, Carter G, Werler M, Jones H. Naltrexone Treatment for Pregnant Women With Opioid Use Disorder Compared With Matched Buprenorphine Control Subjects. Clin Ther. 2019 Sep;41(9):1681-1689. doi: 10.1016/j.clinthera.2019.07.003. Epub 2019 Jul 27. PMID 31358302